CLINICAL TRIAL: NCT04747912
Title: A Phase II Study of a Chemotherapy-Free Induction Regimen for Ph+ Acute Lymphoblastic Leukemia (ALL) Incorporating Inotuzumab Ozogamicin (InO)
Brief Title: Study of Chemotherapy-Free Induction Regimen for Ph+ Acute Lymphoblastic Leukemia With Inotuzumab Ozogamicin (InO)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-1749
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia; ph+ Acute Lymphoblastic Leukemia
Keywords: leukemia; Acute Lymphoblastic Leukemia; ph+ Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Inotuzumab Ozogamicin; Dasatinib; Dexamethasone; Calcium Dobesilate; Methotrexate; Vincristine; ponatinib; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm - Induction/Consolidation Phase - All Participants (Experimental): All participants in this arm will receive the same first round of treatment as part of induction/consolidation therapy. This treatment will use inotuzumab ozogamicin combined with anti-cancer drugs. The additional treatment that participants receive after this first round of treatment will vary based on the participant's response to induction therapy. This phase of treatment will last for 60 days. All participants in this arm will receive the following treatment:
  Treatment Course I (Induction Phase, 28 days):
  * Dasatinib 140mg daily continuous
  * Dexamethasone 10mg/m^2 PO or IV Days 1-7 and Day 15-Day 22
  * InO 0.8mg/m2 Day 8; 0.5mg/m2 D15, 0.5mg/m2 Day 22
  * Intrathecal methotrexate 15mg Day 1, Day 28
  Treatment Course II (Consolidation Phase, 28 days):
  * Dasatinib 140mg daily continuous
  * InO: If in CR/CRi 0.5mg/m2 Day 1, Day 8, Day 15; If not in CR/CRi 0.8mg/m2 on Day 1, 0.5mg/m2 Day 8 and Day 15
  * Intrathecal methotrexate 15mg Day 1, Day 28
  Interventions: Drug: Inotuzumab ozogamicin; Drug: Dasatinib; Drug: Dexamethasone; Drug: Methotrexate for Injection
- Treatment Arm - Interim/Maintenance Phase - Participants in CMR (Experimental): This study arm is for participants who no longer show any detectable signs of BCR-ABL1 (a cancer-causing gene) in response to the previous phase of induction/consolidation treatment (also known as being in "complete molecular remission" or CMR). Participants in this arm will receive 3 courses of interim/maintenance treatment using dasatinib combined with other anti-cancer drugs. Inotuzumab ozogamicin will be added during the fourth course of treatment. These treatments will be given in 28-day and 84-day cycles.
  If the participant achieves complete molecular remission (no signs of BCR-ABL gene) after 60 days (or more) of treatment, then the treating physician may take the participant off the study for allogenic stem cell transplantation surgery.
  If the participant does not undergo allogeneic stem cell transplantation after achieving complete molecular remission, they will complete 3 additional courses of maintenance treatment.
  Interventions: Drug: Inotuzumab ozogamicin; Drug: Dasatinib; Drug: Dexamethasone; Drug: Methotrexate; Drug: Vincristine; Drug: Methotrexate for Injection; Procedure: Allogenic Stem Cell Transplantation
- Treatment Arm - Interim/Maintenance Phase - Participants Not in CMR (Experimental): This study arm is for participants whose cancer responded to induction/consolidation treatment, but still shows detectable signs of BCR-ABL1 (a cancer-causing gene), so they are not in complete molecular remission. Participants in this arm will receive 3 courses of treatment using ponatinib combined with other anti-cancer drugs. Inotuzumab ozogamicin will be added during the 4th treatment course. These treatments will be given in 28-day and 84-day cycles.
  If the participant achieves complete molecular remission (no signs of BCR-ABL gene) after 60 days (or more) of treatment, the treating physician may take the participant off the study for allogenic stem cell transplantation surgery.
  If the participant does not undergo allogeneic stem cell transplantation after achieving complete molecular remission (CMR), they will complete 3 additional courses of maintenance treatment.
  If the participant doesn't achieve CMR after 4th treatment course, they will be removed from the study.
  Interventions: Drug: Inotuzumab ozogamicin; Drug: Dexamethasone; Drug: Methotrexate; Drug: Vincristine; Drug: Ponatinib; Drug: Methotrexate for Injection; Procedure: Allogenic Stem Cell Transplantation

INTERVENTIONS:
Drug: Inotuzumab ozogamicin — Inotuzumab ozogamicin, sold under the brand name Besponsa, is an anti-cancer drug used to treat relapsed or refractory B-cell precursor acute lymphoblastic leukemia.
  Other Names: Besponsa
Drug: Dasatinib — Dasatinib is a prescription treatment for adults with newly diagnosed Philadelphia chromosome-positive chronic myeloid leukemia (Ph+ CML).
  Other Names: SPRYCEL
  Arms: Treatment Arm - Induction/Consolidation Phase - All Participants; Treatment Arm - Interim/Maintenance Phase - Participants in CMR
Drug: Dexamethasone — Dexamethasone is a steroid that prevents the release of substances in the body that cause inflammation.
  Other Names: Decadron®, Dexamethasone Intensol®, Dexasone, Solurex®, and Baycadron®
Drug: Methotrexate — Methotrexate is a chemotherapy drug that is used to treat certain types of cancer and leukemia.
  Other Names: Otrexup™, Rasuvo®, Rheumatrex® and Trexall™. MTX, Amethopterin, and Methotrexate Sodium
  Arms: Treatment Arm - Interim/Maintenance Phase - Participants Not in CMR; Treatment Arm - Interim/Maintenance Phase - Participants in CMR
Drug: Vincristine — Vincristine, also known as leurocristine and marketed under the brand name Oncovin among others, is a chemotherapy medication used to treat various types of cancer such as acute lymphocytic leukemia, acute myeloid leukemia, Hodgkin's disease, neuroblastoma, and small cell lung cancer among others.
  Other Names: Oncovin and Vincasar Pfs
  Arms: Treatment Arm - Interim/Maintenance Phase - Participants Not in CMR; Treatment Arm - Interim/Maintenance Phase - Participants in CMR
Drug: Ponatinib — A drug used to treat chronic myelogenous leukemia (CML) and Philadelphia chromosome-positive acute lymphoblastic leukemia. It is used in patients whose cancer has the T315I mutation or whose cancer cannot be treated with other tyrosine kinase inhibitors. It is also being studied in the treatment of other types of cancer. Ponatinib blocks BCR-ABL, which may help keep cancer cells from growing and may kill them.
  Other Names: Iclusig
  Arms: Treatment Arm - Interim/Maintenance Phase - Participants Not in CMR
Drug: Methotrexate for Injection — Methotrexate is a chemotherapy drug that is used to treat certain types of cancer and leukemia. When given intrathecally, it prevents leukemia cells entering the cerebrospinal fluid (CSF) around the spine and brain. Intrathecal chemotherapy is administered during a procedure called a lumbar puncture or through an ommaya reservoir (shunt).
  Other Names: Otrexup™, Rasuvo®, Rheumatrex® and Trexall™. MTX, Amethopterin, and Methotrexate Sodium
Procedure: Allogenic Stem Cell Transplantation — A procedure in which a patient receives healthy blood-forming cells (stem cells) from a donor to replace their own stem cells that have been destroyed by treatment with radiation or high doses of chemotherapy. In an allogeneic stem cell transplant, the healthy stem cells may come from the blood or bone marrow of a related donor who is not an identical twin of the patient or from an unrelated donor who is genetically similar to the patient. An allogeneic stem cell transplant is most often used to treat blood cancers, such as leukemia and lymphoma, and certain types of blood or immune system disorders.
  Arms: Treatment Arm - Interim/Maintenance Phase - Participants Not in CMR; Treatment Arm - Interim/Maintenance Phase - Participants in CMR

SUMMARY:
This research study will add an anti-cancer drug (called inotuzumab ozogamicin also known as "InO") to treatment for participants with newly diagnosed Philadelphia chromosome-positive (Ph+) acute lymphoblastic leukemia (ALL). Doctors leading this study hope to learn if adding InO to standard induction treatment for Ph+ ALL will lead to quicker, complete molecular remission (where the disease is not detectable even with very sensitive testing techniques). The purpose of this research is to gather information regarding the effectiveness of InO in newly-diagnosed Ph+ ALL patients that have not yet received treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a newly diagnosed and untreated patient with Ph+ B-cell Acute Lymphoblastic Leukemia and CD22 expression on ≥20% of blasts.
2. 18 years old or older.
3. Bone marrow involvement with ≥20% lymphoblasts and demonstration of BCR-ABL1 via fluorescence in situ hybridization (FISH) studies or PCR-based testing. Patients with >1000/mm3 lymphoblasts in the peripheral blood that cannot undergo bone marrow biopsy and aspiration due to clinical condition are also eligible.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. Adequate organ function as confirmed by clinical/medical record.
6. Patients must be at least 2 weeks from major surgery, radiation therapy, or participation in other investigational trials, and must have recovered from clinically significant toxicities related to these prior treatments.
7. Patients must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee/Institutional Review Board prior to starting any screening or study-specific procedures.
8. Females of childbearing potential will use effective contraception during treatment with InO and for at least 8 months after the last dose. Males with female partners of reproductive potential will use effective contraception during treatment with Inotuzumab Ozogamicin and for at least 5 months after the last dose. A patient is of childbearing potential if, in the opinion of the treating investigator, he/she is biologically capable of having children and is sexually active. Female patients who are not of childbearing potential (ie, meet at least one of the following criteria):

   a. Have undergone hysterectomy or bilateral oophorectomy; or have medically confirmed ovarian failure; or are medically confirmed to be post-menopausal (cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause).
9. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Isolated extramedullary disease.
2. Burkitt's or mixed-lineage leukemia.
3. Active central nervous system (CNS) leukemia.
4. Any prior therapy for ALL except for limited treatment (≤ 7 days) with corticosteroids or hydroxyurea and a single dose of intrathecal therapy. Patients who are being treated with chronic steroids for other reasons (eg, asthma, autoimmune disorders) are eligible.
5. Current or chronic hepatitis B or C infection as evidenced by hepatitis B surface antigen and anti-hepatitis C antibody positivity, respectively, or known seropositivity for human immunodeficiency virus (HIV). HIV testing may need to be performed in accordance with local regulations or local practice. Patients with HIV but an undetectable viral load are eligible for enrollment
6. Major surgery within ≤ 2 weeks before randomization.
7. Unstable or severe uncontrolled medical condition (eg, unstable cardiac function or unstable pulmonary condition.
8. Concurrent active malignancy other than non-melanoma skin cancer, carcinoma in situ of the cervix, or localized prostate cancer that has been definitely treated with radiation or surgery. Patients with previous malignancies are eligible provided that they have been disease free for ≥2 years or are not currently requiring treatment.
9. Uncontrolled cardiac disease.
10. QTcF > 500 msec (based on the average of 3 consecutive ECGs).
11. History of chronic liver disease (eg, cirrhosis) or suspected alcohol abuse.
12. History of hepatic veno-occlusive disease (VOD) or sinusoidal obstruction syndrome (SOS).
13. Evidence of uncontrolled current serious active infection including sepsis, bacteremia, fungemia, or patients with a recent history (within 4 months) of deep tissue infections such as fasciitis or osteomyelitis.
14. Medications known to predispose to Torsades de Pointes are prohibited throughout the treatment period of the study.
15. Pregnant females; breastfeeding females; males with female partners of reproductive potential and females of childbearing potential not using highly effective contraception or not agreeing to continue highly effective contraception for a minimum of 5 months after the last dose of investigational product if male and 8 months after the last dose of investigational product if female.
16. Patients who are investigational site staff members or relatives of those site staff members or patients who are Pfizer employees directly involved in the conduct of the trial.
17. Participation in other investigational studies during active treatment phase.
18. Other severe acute, chronic medical, psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Study Lead Principal Investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Enter Complete Clinical Remission at 60 Days as Defined by Criteria Set By The International Scale | 60 days
  Complete clinical remission (when there are no signs of the disease) with a major molecular remission at 60 days as defined by participants who have a low ratio (less than or equal to .01%) of BCR-ABL1gene in their blood, according to criteria set by the International Scale for p210 BCR-ABL1.

SECONDARY OUTCOMES:
Overall Survival | 36 months
  The length of time from when the participant first receives study treatment to their death (due to any cause) as assessed by the treating investigator. Participants will be followed for 12 weeks after the last dose of study drug, until any study treatment-related toxicities have stabilized, or until death.
Duration of Response | 36 months
  The length of time from the first documented complete response (participant shows no signs of cancer) or partial response (participant shows fewer signs of cancer) to disease progression or death. Partial/complete response will be assessed by bone marrow biopsies and blood tests.
Duration of Complete Response | 36 months
  The length of time from the first documented complete response (when participant shows no signs of cancer) to disease progression or death as assessed by the treating investigator.
Progression Free Survival | 36 months
  The time from treatment administration to documented disease progression or death from any cause as assessed by the treating investigator.
Disease Control Rate Based on Number of Participants Who Respond to Treatment After 3 Months | 36 months
  The disease control rate based on the number of participants who show a complete response, partial response or no changes in disease (stable disease) after 3 months as assessed by bone marrow biopsies and neutrophil/complete blood count tests.
Number of Participants with Complete Molecular Remission at 180 Days | 36 months
  Number of participants with complete molecular remission at 180 days as defined by the absence of a detectable BCR-ABL1 gene, according to criteria set by the International Scale for p210 BCR-ABL1. Complete molecular remission at 180 days will be assessed among participants who do not undergo allogenic stem cell transplantation after treatment.
Number of Participants With Documented Veno-Occlusive Disease After Treatment | 36 months
  The number of patients with documented veno-occlusive disease as assessed by treating investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States